CLINICAL TRIAL: NCT01598831
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Assess the Safety and Efficacy of ART-123 in Subjects With Severe Sepsis and Coagulopathy.
Brief Title: Phase 3 Safety and Efficacy Study of ART-123 in Subjects With Severe Sepsis and Coagulopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asahi Kasei Pharma America Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3-001
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-03

CONDITIONS: Severe Sepsis; Coagulopathy
Keywords: sepsis
MeSH Terms: conditions — Sepsis; Hemostatic Disorders | interventions — ART123

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ART-123 (Active Comparator)
  Interventions: Drug: ART-123
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ART-123 — Dose: 0.06 mg/kg/day up to a maximum dose of 6 mg/day for 6 days
  Other Names: human recombinant thrombomodulin; thrombomodulin alfa
  Arms: ART-123
Drug: Placebo — Dose: 0.06 mg/kg/day up to a maximum dose of 6 mg/day for 6 days.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate if ART-123 given to patients who have severe sepsis can decrease mortality.

DETAILED DESCRIPTION:
Study is to evaluate if ART-123 given to patients who have severe sepsis complicated by at least one organ dysfunction and coagulopathy can decrease mortality.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be receiving treatment in an ICU, or in an acute care setting (e.g., ER, RR)
* Clinical objective evidence of bacterial infection and a known site of infection.
* Cardiovascular dysfunction or Respiratory Failure due to sepsis.
* Coagulopathy characterized by an INR >1.40 without other known causes.

Exclusion Criteria:

* Subject or Authorized Representative is unable to provide informed consent.
* Subject is pregnant or breastfeeding or intends to get pregnant within 28 days of enrolling into the study.
* Subject is of childbearing potential and does not have a negative pregnancy test.
* Subject is < 18 years of age.
* Subject has a known allergy to ART-123 or any components of the drug product.
* Subject is unwilling to allow transfusion of blood or blood products.
* Subject has an advance directive to withhold life-sustaining treatment.
* Subject has had previous treatment with ART-123.
* Body weight ≥ 175 kg.
* Platelets < 30,000/ mm3 for any reason, PT prolongation or thrombocytopenia that is not due to sepsis.
* Any surgery that is potentially hemorrhagic (e.g. intra-thoracic, intra-abdominal or non-traumatic orthopedic surgery of the femur or pelvis) that is completed within 12 hours prior to first dose of study drug, or ongoing impairment of hemostasis as a result of one of these procedures
* History of head trauma, spinal trauma, or other acute trauma with an increased risk of bleeding within 3 months prior to consent.
* Cerebral Vascular Accident (CVA) within 3 months prior to consent.
* Any history of intracerebral arteriovenous malformation (AVM), cerebral aneurysm, or mass lesions of the central nervous system.
* History of congenital bleeding diathesesor anatomical anomaly that predisposes to hemorrhage (e.g. hemophilia, hereditary hemorrhagic telangiectasia).
* Significant gastrointestinal bleeding within 6 weeks prior to consent.
* Subject is diagnosed with a known medical condition associated with a hypercoagulable state.
* Child-Pugh score of 10-15 (Class C)
* Portosystemic hypertension or known history of bleeding esophageal varices.
* History of solid organ, allogeneic bone marrow, or stem cell transplantation within the 6 months prior to consent.
* Acute pancreatitis where infection has not been documented by a positive blood or abdominal fluid culture or gram stain consistent with bacterial infection.
* Subjects with renal dysfunction defined as (a) Chronic renal failure requiring renal replacement therapy (RRT), or (b) Acute renal failure with onset of oliguria (urine output < 0.3 ml/kg/hr) > 48 hours prior to first dose of study drug whether receiving RRT or not
* Use of anticoagulants, antiplatelet agents, antithrombotics and thrombolytics within the 72 hours prior to first does of study drug.
* Life expectancy < 90 days.
* Current use of any chemotherapy agent likely to cause myeloablation (severe or complete depletion of bone marrow).
* Participation in another research study involving an investigational agent within 30 days prior to consent or projected study participation during the 28 days post study randomization.
* Confirmed or suspected endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 816 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Fineberg, M.D., Study Director — Asahi Kasei Pharma America Corporation
Locations (160):
- United States (22):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Atlanta, Georgia
  - Idaho Falls, Idaho
  - Indianapolis, Indiana
  - Hazard, Kentucky
  - Louisville, Kentucky
  - Detroit Receiving Hospital, Detroit, Michigan
  - Harper Hospital - Wayne State University School of Medicine, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - Jackson, Mississippi
  - Washington University in St. Louis, St Louis, Missouri
  - Butte, Montana
  - Englewood, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Durham, North Carolina
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Rapid City, South Dakota
  - 2 of 2, Houston, Texas
  - Murray, Utah
- Hospital Italiano de Cordoba, Córdoba, Argentina
- Australia (10):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Bendigo Hospital, Bendigo, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Dandenong Hospital Monash Health, Dandenong, Victoria
  - Western Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Sunshine Hospital, Melbourne, Victoria
- Belgium (11):
  - UZ Antwerpen, Antwerp
  - Cliniques Du Sud-Luxerbourg (CSL), Hospital Saint Joseph, Arlon
  - CHU Brugmann, Brussels
  - Hopital Erasme, Brussels
  - Hopitaux Iris Sud, Brussels
  - UCL St. Luc, Brussels
  - UZ Brussel, Brussels
  - Centre Hospitalier de Dinant, Dinant
  - UZ Gent, Ghent
  - Clinique Saint-Pierre, Ottignies
  - UCL Mont-Godinne, Yvoir
- Brazil (3):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Fundaçao Faculdade Regional de Medicina Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Pompéia, Brasil
- Bulgaria (2):
  - Anesthesiology and Intensive Care Clinic, University Multiprofile Hospital For Active Treatment "Sveti Georgi", Plovdiv, Plovdiv
  - Department of Anesthesiology and Intensive Care Multiprofile Hospital For Active Treatment "Tokuda Hospital Sofia", Sofia, Sofia
- Canada (13):
  - 2 of 2, Calgary, Alberta
  - Calgary, Alberta
  - Vancouver, British Columbia
  - 2 of 2, Vancouver, British Columbia
  - 1 of 2, Victoria, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
  - 1 of 2, Ottawa, Ontario
  - 2 of 2, Ottawa, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
- Croatia (3):
  - Clinical Hospital Center Zagreb, Medical ICU, Zagreb
  - Clinical Hospital Dubrava, Department of Anesthesiology and resuscitation, Zagreb
  - University Hospital Center Zagreb, Department of Anesthesiology, Reanimatology and Intensive Care Medicine, Zagreb
- Czechia (5):
  - University Hospital Brno, Department of Infectious Diseases, Brno
  - University Hospital Hradec Kralove, Department of Anaesthesiology, Resuscitation and Intensive Care, Hradec Králové
  - General University Hospital in Prague, Department of Anaesthesiology, Resuscitation and Intensive Medicine, Prague
  - University Hospital Kralovske Vinohrady, Department of Anesthesiology and Resuscitation, Prague
  - Masaryk´s Hospital Ustni nad Labem, o.z., Department of Infectious Diseases, Ústí nad Labem
- Finland (4):
  - Helsingin Yliopistollinen Keskussairaala (HYKS) (Helsinki University Central Hospital (HUCH)), Helsinki
  - Keski-Suomen Keskussairaala (Central Finland Central Hospital), Jyväskylä
  - Kuopion Yliopistollinen Sairaala (KYS) (Kuopio University Hospital), Kuopio
  - Tampereen Yliopistollinen Sairaala (Tampere University Hospital) (TAYS) - Keskussairaala (Central Hospital), Tampere
- France (16):
  - Archet 1 University Hospital of Nice, Nice, Cedex 3
  - Service de reanimation médicale. CHU Hotel Dieu, Nantes, Nantes Cedex 01
  - CHU D'Anger, Angers
  - CHU de Dijon, Hopital Bocage Central, Dijon
  - CH-Hôpital Albert Michallon, Grenoble
  - Centre Hospitalier Départemental de Vendée-Les Oudairies, La Roche-sur-Yon
  - CHRU Lille-Pole Reanimation, Lille
  - CHU Limoges, Limoges
  - Centre Hospitalier Universitaire Nîmes, Nîmes
  - La Pitié Salpétrière, Paris, Paris
  - Hôpital COCHIN, Paris
  - University Hospital of Bordeaux, Pessac
  - CH Lyon Sud, Pierre-Bénite
  - Nouvel hospital civil, Strasbourg
  - Hôpital Sainte Musse, Toulon
  - CHU Tours, Hopital Bretonneau, Tours
- Germany (3):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Helios Klinikum Erfurt, Erfurt
  - Klinikum der Johann-Wolfgang Goethe-Universität, Frankfurt am Main
- Szent Imre Hospital, Anesthesiology and Intensive Care Unit, Budapest, Hungary
- India (15):
  - Shalby Hospital, Ahmedabad, Gujarat
  - Shalby, Ahmedabad, Gujarat
  - Artemis Hospital, Gurgaon, Haryana
  - Ruby Hall Clinic, Pune, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - King Edward Memorial Hospital & Research Centre, Pune, Maharashtra
  - Maulana Azad Medical College and Associated L N Hospital, New Delhi, National Capital Territory of Delhi
  - Hi-tech Medical College & Hospital, Bhubaneswar, Odisha
  - Bharati Vidyapeeth Deemed University Medical College Bharti Hospital and Research Centre, Pune, Pune, Maharashtra
  - St. Theresa Hospital, Hyderabad, Telangana State
  - Mazumdar Shaw Medical Centre (Unit of Narayana Health), Bangalore
  - KLES Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi
  - JSS Hospital, Mysore
  - Care Hospital, Nagpur
  - Noble Hospital, Pune
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Netherlands (8):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - VUMC, Amsterdam
  - Ziekenhuis Gelderse Vallei, Ede
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - UMC St. Radboud, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
- New Zealand (4):
  - Auckland District Health Board, Auckland
  - Christchurch Hospital, Christchurch
  - Hawkes Bay Regional Hospital Intensive Care Unit Omahu Road, Hastings
  - Wellington District Health Board, Newtown
- Peru (2):
  - Hospital Nacional Almenara Yrigoyen - EsSALUD, Lima, Lima Province
  - Hospital Nacional FAP, Lima, Lima Province
- Russia (12):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Volosevich City Clinical Hospital #1, Arkhangelsk
  - City Clinical Hospital #3 n.a. M.A. Pogorbunskiy, Kemerovo
  - Kuban State Medical University (Site Facility: Krasnodar Regional Clinical Hospital #2), Krasnodar
  - Krasnoyarsk Regional Clinocal Hospital, Krasnoyarsk
  - Vishnevsky Institute of Surgery, Moscow
  - St George City Hospital, Saint Petersburg
  - Aleksandrovskaya City Hospital, Saint Petersburg
  - City Hospital #40, Saint Petersburg
  - Mariinskaya City Hospital, Saint Petersburg
  - Mechnikov North-Western State Medical University n.a. I.I. Mechnikov, Saint Petersburg
  - City Hospital #4, Sochi
- Clinic for Infectious Diseases, Clinical Center Nis, Niš, Serbia
- South Korea (4):
  - Korea University Anam Hospital, Seongdu
  - Asan Medical Center, Seoul
  - Samsung Medical Center [Pulmonology], Seoul
  - Seoul National University Hospital, Seoul
- Spain (6):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Mutua Terrassa Intensive Care, Barcelona
  - Servicio de Medicina Intensiva Hospital Universitario Valle de Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital de Sabadell, Sabadell
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona
- Taiwan (3):
  - Chi Mei Medical Center Yong Kang, Yongkang District, Tainan
  - Taichung Veterans General Hospital [Pulmonology], Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - Hull Royal Infirmary, Hull
  - Royal Liverpool University Hospital, Liverpool
  - Manchester Royal Infirmary, Manchester
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Levi M, Vincent JL, Tanaka K, Radford AH, Kayanoki T, Fineberg DA, Hoppensteadt D, Fareed J. Effect of a Recombinant Human Soluble Thrombomodulin on Baseline Coagulation Biomarker Levels and Mortality Outcome in Patients With Sepsis-Associated Coagulopathy. Crit Care Med. 2020 Aug;48(8):1140-1147. doi: 10.1097/CCM.0000000000004426. PMID 32697484
- [Derived] Vincent JL, Francois B, Zabolotskikh I, Daga MK, Lascarrou JB, Kirov MY, Pettila V, Wittebole X, Meziani F, Mercier E, Lobo SM, Barie PS, Crowther M, Esmon CT, Fareed J, Gando S, Gorelick KJ, Levi M, Mira JP, Opal SM, Parrillo J, Russell JA, Saito H, Tsuruta K, Sakai T, Fineberg D; SCARLET Trial Group. Effect of a Recombinant Human Soluble Thrombomodulin on Mortality in Patients With Sepsis-Associated Coagulopathy: The SCARLET Randomized Clinical Trial. JAMA. 2019 May 28;321(20):1993-2002. doi: 10.1001/jama.2019.5358. PMID 31104069
- See also: Information on sepsis and treatment — http://internationalsepsisforum.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 319 sites in 27 countries; of these, 159 study sites (in 26 countries) assigned participants to study drug treatment. First participant was randomized on Oct 29, 2012 and the last participant was randomized on Mar 8, 2018. Last participant completed long term follow-up (survival only) on Feb 28, 2019.
Pre-assignment Details: Of 946 consented participants, 816 randomized to study treatment, 800 received at least 1 dose of study treatment.
Groups:
- ART-123: ART-123 (human recombinant thrombomodulin, thrombomodulin alfa) Dose: 0.06 mg/kg/day up to a maximum dose of 6 mg/day for 6 days
- Placebo: Placebo Dose: 0.06 mg/kg/day up to a maximum dose of 6 mg/day for 6 days
Period: Overall Study
Arm/Group | ART-123 | Placebo
Started | 402 | 414
Received at Least 1 Dose Study Treatment | 395 | 405
Completed | 283 | 278
Not Completed | 119 | 136

BASELINE CHARACTERISTICS:
Population: Baseline characteristic is an overview of participants who received at least one dose (Full Analysis Set)
Groups:
- Total: Total of all reporting groups
Arm/Group | ART-123 | Placebo | Total
Number analyzed (Participants) | 395 | 405 | 800
Age, Categorical [Count of Participants; unit: Participants] — Count of participants in each age group at baseline
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 231 | 231 | 462
    >=65 years | 164 | 174 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants Age in years (Mean, SD) at baseline
  years | 61.0 (15.87) | 60.5 (15.94) | 60.7 (15.89)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants Sex at baseline
  Participants
    Female | 179 | 184 | 363
    Male | 216 | 221 | 437
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants ethnicity at baseline
  Participants
    Hispanic or Latino | 20 | 22 | 42
    Not Hispanic or Latino | 290 | 285 | 575
    Unknown or Not Reported | 85 | 98 | 183
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants race at baseline
  Participants
    American Indian or Alaska Native | 5 | 8 | 13
    Asian | 56 | 58 | 114
    Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
    Black or African American | 14 | 20 | 34
    White | 312 | 308 | 620
    More than one race | 7 | 9 | 16
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Number of participants enrolled by country
  Participants
    United States | 34 | 37 | 71
    Czechia | 10 | 11 | 21
    Russia | 54 | 57 | 111
    Greece | 0 | 1 | 1
    Netherlands | 22 | 27 | 49
    South Korea | 4 | 2 | 6
    Brazil | 11 | 8 | 19
    Bulgaria | 1 | 1 | 2
    France | 75 | 74 | 149
    Serbia | 1 | 1 | 2
    Croatia | 6 | 5 | 11
    Colombia | 2 | 0 | 2
    Argentina | 1 | 0 | 1
    Hungary | 0 | 1 | 1
    United Kingdom | 6 | 4 | 10
    India | 41 | 44 | 85
    Spain | 9 | 11 | 20
    New Zealand | 6 | 5 | 11
    Canada | 22 | 24 | 46
    Belgium | 34 | 34 | 68
    Finland | 18 | 19 | 37
    Taiwan | 4 | 4 | 8
    Israel | 9 | 10 | 19
    Australia | 19 | 19 | 38
    Peru | 3 | 2 | 5
    Germany | 3 | 4 | 7
Height [Mean (Standard Deviation); unit: cm] — Participant Height (mean, SD) Population: One subject in the ART-123 arm and one in the Placebo arm did not have baseline height recorded in the eCRF
  cm
    number analyzed (Participants) | 394 | 404 | 798
    (all) | 167.39 (8.729) | 168.02 (9.619) | 167.71 (9.190)
Weight [Mean (Standard Deviation); unit: kg] — Participant Weight (mean, SD) Population: One subject in the ART-123 arm did not have baseline weight recorded in the eCRF
  kg
    number analyzed (Participants) | 394 | 405 | 799
    (all) | 75.01 (19.131) | 75.74 (19.266) | 75.38 (19.191)
APACHE II (mean, SD) [Mean (Standard Deviation); unit: Total Score] — APACHE II is a scoring system to grade the severity of illness in critically ill patients that generates a score based on age and 12 physiologic variables of underlying health (Temperature, Mean arterial pressure, Heart rate, Respiratory rate, Oxygenation, Arterial pH, Serum sodium, Serum potassium, Serum creatinine, Hematocrit, WBC, Glasgow coma score). Total APACHE II score = sum of the 12 individual variable points +age points + chronic health points. Min score = 0; Max score = 71. Increasing score is associated with increasing risk of hospital death. Population: Subjects in the ART-123 and Placebo arms did not have baseline Apache II recorded in the eCRF
  Total Score
    number analyzed (Participants) | 356 | 366 | 722
    (all) | 22.34 (8.071) | 22.10 (8.025) | 22.22 (8.043)
Arterial Lactate >55mg/dl (mean, SD) [Count of Participants; unit: Participants] — Patients with septic shock can be clinically identified by a vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia (Singer 2016 JAMA). Further increase in the levels of lactate are a marker of even higher illness severity and 55 mg/dL was selected as a measure of very high illness severity' Population: Subjects in the ART-123 and Placebo arms did not have baseline Arterial Lactate recorded in the eCRF
  Participants
    number analyzed (Participants) | 253 | 279 | 532
    (all) | 53 | 52 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 28-Day All-cause Mortality
Description: 28-Day All-cause Mortality
Time Frame: 28 days
Population: Full Analysis Set - All randomized and dosed subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | ART-123 | Placebo
Number analyzed (Participants) | 395 | 405
Participants | 106 | 119
Statistical Analysis 1: Comparison: ART-123 vs Placebo; Test type: Superiority; p = 0.318, Cochran-Mantel-Haenszel — The threshold for statistical significance was a two sided 5%; CMH test controlled for the stratification factor; Risk Difference (RD) = -2.55, 95% CI 2-sided [-3.68 to 8.77] — Rates by Arm are 26.8% for ART-123 and 29.4% for Placebo; In a post hoc sensitivity analysis for the primary outcome that accounted for pooled site as a random effect, the adjusted 28-day all-cause mortality rate was 24.8%in the rhsTM group vs 27.5%in the placebo group (P = .31)

2. Primary Outcome: Number of Participants With On-Treatment Serious Major Bleeding Events
Description: On-treatment Serious Major Bleeding Events collected as Serious Adverse Events and defined as: any intracranial hemorrhage, any life-threatening bleeding, any bleeding event classified as serious by the Investigator (e.g., resulting in permanent morbidity), or any bleeding that required the administration of 1440 ml (typically 6 units) of packed red cells over two consecutive days. (Investigator assessment for seriousness criteria.)
Time Frame: Through Study Day 28
Population: Safety population: all subjects who received at least 1 dose of study drug (analyzed according to study drug received; any subjects receiving both ART-123 and placebo were to be included in the ART-123 group)
Measure: Count of Participants; unit: Participants
Arm/Group | ART-123 | Placebo
Number analyzed (Participants) | 396 | 404
Participants | 23 | 16

3. Secondary Outcome: Follow up All-cause Mortality at 3 Months
Description: Follow up all-cause mortality at 3 months
Time Frame: 3 months
Population: Full Analysis Set - All randomized and dosed subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | ART-123 | Placebo
Number analyzed (Participants) | 395 | 405
Participants | 126 | 136

4. Secondary Outcome: Number of Event Free and Alive Days to Measure Resolution of Organ Dysfunction
Description: Resolution of organ dysfunction as measured through day 28 by shock free, ventilator free, dialysis free plus alive days.
Time Frame: 28 days
Population: Full Analysis Set - All randomized and dosed subjects.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ART-123 | Placebo
Number analyzed (Participants) | 395 | 405
Days
  Shock-free and alive | 17.6 (10.50) | 17.6 (10.56)
  Ventilation-free and alive | 15.8 (11.75) | 14.5 (11.90)
  Dialysis-free and alive | 20.2 (11.05) | 19.6 (11.21)

5. Secondary Outcome: Number of Participants With Anti-drug Antibodies
Description: Presence of Anti-drug antibodies up to 18 months
Time Frame: 18 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ART-123 | Placebo
Number analyzed (Participants) | 396 | 404
Participants | 0 | 0

6. Post Hoc Outcome: Day 28 Mortality in Subjects With INR > 1.4 at Baseline and PLT > 30K at Baseline
Description: Post-Hoc analysis of Day 28 Mortality in Subjects with INR > 1.4 at Baseline and PLT > 30K at Baseline
Time Frame: Day 28
Population: Full Analysis Set - All randomized and dosed subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | ART-123 | Placebo
Number analyzed (Participants) | 307 | 327
Participants | 82 | 105

ADVERSE EVENTS:
Time Frame: Adverse events were collected between randomization and through Day 28 only. SAEs were collected from the time of authorization to randomize the participants until Day 28. All-cause mortality were collected as Fatal SAEs between randomization and Day 28 (End of Study) and as survival follow-up from Day 28 until 12 months.
Description: AEs were analyzed using a safety population that includes all subjects who received at least 1 dose of study drug (analyzed according to study drug received; any subjects receiving both ART-123 and placebo were to be included in the ART-123 group). Treatment Emergent Serious Adverse Events (TESAE) were analyzed by System Organ Class and Preferred Term. A treatment-emergent adverse event (TEAE) is defined as any AE following exposure to study treatment.
Arm/Group | ART-123 | Placebo
All-Cause Mortality (participants affected / at risk) | 141/395 | 148/405
Serious Adverse Events (participants affected / at risk) | 206/396 | 202/404
Other Adverse Events (participants affected / at risk) | 271/396 | 264/404
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ART-123 (N=396) | Placebo (N=404)
Septic shock (Infections and infestations) | 28 | 30
Sepsis (Infections and infestations) | 8 | 11
Pneumonia (Infections and infestations) | 8 | 10
Peritonitis (Infections and infestations) | 3 | 3
Gangrene (Infections and infestations) | 3 | 2
Necrotising fasciitis (Infections and infestations) | 1 | 3
Endocarditis (Infections and infestations) | 2 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 1
Abdominal sepsis (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cellulitis gangrenous (Infections and infestations) | 0 | 1
Fungal sepsis (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0
Herpes simplex pneumonia (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Infective aneurysm (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 1 | 0
Septic embolus (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Varicella zoster pneumonia (Infections and infestations) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragm muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 10 | 11
Atrial fibrillation (Cardiac disorders) | 6 | 5
Bradycardia (Cardiac disorders) | 4 | 2
Cardiac failure acute (Cardiac disorders) | 4 | 2
Cardiopulmonary failure (Cardiac disorders) | 2 | 3
Myocardial infarction (Cardiac disorders) | 1 | 3
Cardio-respiratory arrest (Cardiac disorders) | 3 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 24 | 28
Death (General disorders) | 0 | 2
Pyrexia (General disorders) | 2 | 0
Catheter site haematoma (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1
Organ failure (General disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 7 | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 5
Gastrointestinal necrosis (Gastrointestinal disorders) | 3 | 2
Intestinal perforation (Gastrointestinal disorders) | 3 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Fistula of small intestine (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal wall abnormal (Gastrointestinal disorders) | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Mesenteric haemorrhage (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 6 | 6
Shock (Vascular disorders) | 4 | 7
Deep vein thrombosis (Vascular disorders) | 2 | 4
Shock haemorrhagic (Vascular disorders) | 6 | 0
Hypotension (Vascular disorders) | 1 | 2
Arterial occlusive disease (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 1
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 14 | 10
Renal failure (Renal and urinary disorders) | 3 | 1
Renal impairment (Renal and urinary disorders) | 2 | 1
Anuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal ischaemia (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 12
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 6 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 4
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 2
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 4 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2
Embolic cerebral infarction (Nervous system disorders) | 2 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 1
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 2
Brain hypoxia (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 0 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hypercapnic coma (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 3
Hepatocellular injury (Hepatobiliary disorders) | 2 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0
Platelet count decreased (Investigations) | 2 | 0
Coma scale abnormal (Investigations) | 1 | 0
Glutamate dehydrogenase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
International normalised ratio abnormal (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1
Adrenal haemorrhage (Endocrine disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ART-123 (N=396) | Placebo (N=404)
Anaemia (Blood and lymphatic system disorders) | 99 | 78
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 51
Atrial fibrillation (Cardiac disorders) | 51 | 52
Constipation (Gastrointestinal disorders) | 37 | 37
Diarrhoea (Gastrointestinal disorders) | 31 | 36
Nausea (Gastrointestinal disorders) | 31 | 18
Pyrexia (General disorders) | 39 | 33
Oedema peripheral (General disorders) | 20 | 17
Pneumonia (Infections and infestations) | 21 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 83 | 69
Hypophosphataemia (Metabolism and nutrition disorders) | 46 | 39
Hyperglycaemia (Metabolism and nutrition disorders) | 37 | 34
Hypoglycaemia (Metabolism and nutrition disorders) | 25 | 31
Hyperkalaemia (Metabolism and nutrition disorders) | 25 | 20
Hypomagnesaemia (Metabolism and nutrition disorders) | 25 | 19
Hypernatraemia (Metabolism and nutrition disorders) | 21 | 22
Fluid overload (Metabolism and nutrition disorders) | 21 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 21 | 11
Delirium (Psychiatric disorders) | 31 | 21
Insomnia (Psychiatric disorders) | 20 | 21
Acute kidney injury (Renal and urinary disorders) | 28 | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 27 | 31
Hypertension (Vascular disorders) | 23 | 25
Hypotension (Vascular disorders) | 23 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT01598831/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT01598831/SAP_001.pdf